CLINICAL TRIAL: NCT06649734
Title: Consensus Statements on Airway Clearance Interventions in Intubated Critically Ill Patients--Protocol for a Delphi Study
Acronym: ACCorDingly
Status: Not yet recruiting | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: The Royal Wolverhampton Hospitals NHS Trust (Other Government)
Responsible Party: Principal Investigator, Prof. Dr. Marcus J. Schultz, professor dr., Amsterdam University Medical Centers (UMC), Location Academic Medical Center (AMC)
Other Study IDs: ACCorDingly
Record Dates: First submitted 2024-10-01; First posted 2024-10-21 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Critically Ill; Ventilation Therapy; Complications; Mucus Retention; Airway Clearance Impairment
Keywords: Airway Clearance Techniques
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Expert Panel: An international expert panel of at least 35 to 40 healthcare professionals representing ICU-nurses, respiratory therapists (or comparable version, based on local implementation), physiotherapists, ICU-physicians and pulmonologists with expertise in the field of invasively ventilated ICU-patients.
  Interventions: Other: Delphi Study

INTERVENTIONS:
Other: Delphi Study — A Delphi study will be conducted with several rounds up to stable expert consensus or dissensus

SUMMARY:
Intubated critically ill patients are susceptible to secretion accumulation because of compromised airway clearance. Various airway clearance interventions are employed to prevent complication(s) arising from mucus retention. Available guidelines are largely based on clinical expertise and low-level evidence, with no international consensus on their use. This Delphi study aims to collect global opinions on the usefulness of these various airway clearance interventions. Statements are grouped into two distinct parts: (1) Humidification and Nebulization, and (2) Suctioning and Secretion mobilization techniques.

DETAILED DESCRIPTION:
Introduction Intubated critically ill patients are susceptible to secretion accumulation because of compromised airway clearance. Various airway clearance interventions are employed to prevent complication arising from mucus retention. This Delphi study aims to collect global opinions on the usefulness of these various airway clearance interventions. The diverse expertise of the panel will provide valuable insights for refining airway care for intubated critically ill patients, eventually improving outcomes.

Methods The steering committee, comprising of 10 healthcare professionals working in intensive care including two Delphi methodologists, performed a focused literature search on airway clearance methods and drafted statements. Statements are grouped into two distinct parts: (1) Humidification and Nebulization, and (2) Suctioning and Secretion mobilization techniques. For each Delphi part a diverse panel of 35-40 experts will be selected, with concerted effort to involve experts from various medical specialties involved in airway clearance methods inclusive of, but not limited to ICU nurses, respiratory therapists, physiotherapists, intensive care physicians. The identity of these experts will stay anonymized from each other until the end of the Delphi process. Multiple choice questions (MCQs) or 7-point Likert-scale statements will be used in the iterative Delphi rounds to reach consensus on various airway clearance interventions. Comments and feedback from experts will be collected during each Delphi round. Anonymized survey report and comments will be shared with other experts along with link for the consecutive survey. The Delphi rounds will be continued until a stable agreement or disagreement is achieved for all statements. The steering committee will not participate in the voting process during Delphi rounds.

Analysis Consensus will be deemed achieved when a choice in MCQs or a Likert-scale statement achieves ≥ 75% agreement or disagreement. Starting from the second round of the Delphi process, stability will be assessed using non-parametric χ2 tests or Kruskal-Wallis tests. Stability will be defined by a P-value of ≥ 0.05.

Ethics and dissemination The study will be conducted in strict accordance with the principles of the Declaration of Helsinki and reported following ACCORD guidelines. An ethical approval waiver has been granted, due to the nature of the research. Participation in the study is voluntary, and completing and returning the survey will be considered as explicit consent to take part in the study. The study results will be published in a peer-reviewed journal. Patients' representatives will be involved to ensure their perspectives are considered throughout the research process.

ELIGIBILITY:
Healthcare professionals will be selected as panelists based on the following criteria:

Inclusion criteria:

* at least 5 years of clinical experience, with care for invasively ventilated patients (teaching and non-teaching); and
* participation in development of a guideline or authorship of at least one peer reviewed published paper in airway care for invasive ventilated patients; and
* not more than 70% of the panelists from each sex; and from each of high and low- and middle-income countries.

Exclusion criteria:

- none

Purposive sampling will be utilized to recruit panelists by reviewing recent publications in the field of airway care for invasive ventilated patients. Selection of panelists will be guided by predefined criteria, with deliberate efforts to ensure a balance in gender and geographical representation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthcare professionals representing ICU-nurses, respiratory therapists (or comparable version, based on local implementation), physiotherapists, ICU-physicians and pulmonologists with expertise in the field of invasively ventilated ICU patients.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Consensus use of airway clearance intervention Humidification | Time Frame: 3-6 months
  Diverse group of panelist across the globe based on pre-specified qualification criteria and will conduct iterative Delphi rounds to generate consensus on Humidification in invasively ventilated Intensive Care patients.
Consensus use of airway clearance intervention Inhaled Therapy | Time Frame: 3-6 months
  Diverse group of panelist across the globe based on pre-specified qualification criteria and will conduct iterative Delphi rounds to generate consensus on Inhaled Therapy in invasively ventilated Intensive Care patients.
Consensus use of airway clearance intervention Endotracheal Suctioning | Time Frame: 3-6 months
  Diverse group of panelist across the globe based on pre-specified qualification criteria and will conduct iterative Delphi rounds to generate consensus on Endotracheal Suctioning in invasively ventilated Intensive Care patients.
Consensus use of airway clearance intervention Mucus Mobilisation techniques | Time Frame: 3-6 months
  Diverse group of panelist across the globe based on pre-specified qualification criteria and will conduct iterative Delphi rounds to generate consensus on Mucus Mobilisation techniques in invasively ventilated Intensive Care patients.

CONTACTS AND LOCATIONS:
Overall Officials: Frederique Paulus, prof. dr., Principal Investigator — Amsterdam UMC